CLINICAL TRIAL: NCT06500273
Title: A Randomized, Open-label Study Evaluating the Efficacy and Safety of Cemacabtagene Ansegedleucel in Participants With Minimal Residual Disease After Response to First Line Therapy for Large B-cell Lymphoma
Brief Title: Consolidation of First-Line MRD+ Remission With Cema-cel in Patients With LBCL
Acronym: ALPHA3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Allogene Therapeutics (Industry)
Collaborators: Foresight Diagnostics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-501A-202
Record Dates: First submitted 2024-06-26; First posted 2024-07-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Large B-cell Lymphoma
Keywords: Diffuse large B-cell lymphoma; DLBCL; Primary mediastinal B-cell lymphoma; LBCL; High grade B-cell lymphoma; HGBCL; Double-hit lymphoma; High-risk lymphoma; Minimal Residual Disease; MRD; CAR T; Allogeneic CAR T; CD19; cema-cel; cemacabtagene ansegedleucel; PMBCL; Consolidation; First-line; Front-line; Frontline; PhasED-Seq™; CLARITY™; AlloCAR T™
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Neoplasm, Residual | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- cemacabtagene ansegedleucel (Experimental): Participants receive cemacabtagene ansegedleucel following lymphodepletion regimen comprised of fludarabine and cyclophosphamide.
  Interventions: Genetic: cemacabtagene ansegedleucel; Drug: Fludarabine; Drug: Cyclophosphamide; Device: Foresight CLARITY™ IUO MRD test, powered by PhasED-Seq™
- Observation (Other): Participants do not receive any study treatments. They are observed as per the current standard of care.
  Interventions: Device: Foresight CLARITY™ IUO MRD test, powered by PhasED-Seq™

INTERVENTIONS:
Genetic: cemacabtagene ansegedleucel — An allogeneic CAR T cell therapy targeting CD19
  Other Names: cema-cel
  Arms: cemacabtagene ansegedleucel
Drug: Fludarabine — Chemotherapy for lymphodepletion
  Other Names: Fludara®
  Arms: cemacabtagene ansegedleucel
Drug: Cyclophosphamide — Chemotherapy for lymphodepletion
  Other Names: Cytoxan®
  Arms: cemacabtagene ansegedleucel
Device: Foresight CLARITY™ IUO MRD test, powered by PhasED-Seq™ — A diagnostic test intended to identify patients with minimal residual disease at the end of first line treatment for LBCL.
  Other Names: Foresight Lymphoma MRD Therapy Selection Test

SUMMARY:
This is a randomized, open-label study in adult patients who have completed standard first line therapy for large B-cell lymphoma (LBCL) and achieved a complete response or partial response suitable for observation, but who have minimal residual disease (MRD) as detected by the Foresight CLARITY™ Investigational Use Only (IUO) MRD test, powered by PhasED-Seq™. The purpose of the trial is to assess the efficacy and safety of consolidation with cemacabtagene ansegedleucel (cema-cel), an allogeneic CD19 CAR T product, as compared to standard of care observation.

In this study, participants with MRD are randomized 1:1 to treatment with cema-cel or an observation arm. Treatment includes cema-cel following a lymphodepletion regimen of fludarabine and cyclophosphamide.

Prior to August 2025, participants may also have received an anti-CD52 monoclonal antibody, ALLO-647, as part of their lymphodepletion regimen.

ELIGIBILITY:
Key Inclusion Criteria:

1. LBCL per WHO 2017 including diffuse large B-cell lymphoma, high-grade B-cell lymphoma, and primary mediastinal B-cell lymphoma histologically confirmed by pathology report.
2. Participant has completed a full course of standard first line therapy (e.g., R-CHOP, dose-adjusted EPOCH-R, Pola-R-CHP) as intended. Participants cannot have received additional lines of therapy.
3. Participant achieved CR, or PR suitable for observation, at the end of first line therapy based on PET/CT evaluation
4. Foresight CLARITY™ IUO MRD test, powered by PhasED-Seq™, is positive.
5. Adult participants ≥18 years of age.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
7. Adequate hematological, renal, hepatic, pulmonary, and cardiac function
8. Non-hematologic toxicities related to prior therapy must be recovered to baseline or grade ≤1.

Key Exclusion Criteria:

1. LBCL with history of central nervous system involvement, transformed from other malignancy (e.g., transformed follicular lymphoma or marginal zone lymphoma, Richter's transformation), or T-cell/histiocyte rich LBCL.
2. Prior treatment with anti-CD19 targeted therapies.
3. Anti-cancer treatment, including radiation, after end of treatment PET/CT and/or MRD testing is performed.
4. Active and clinically significant autoimmune disease.
5. Active systemic bacterial, fungal, or viral infections requiring systemic treatment.
6. History of another primary malignancy or bone marrow disorder (e.g., myelofibrosis, smoldering multiple myeloma) within 3 years prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-08-24 (Estimated); Study Completion 2031-08-24 (Estimated)

PRIMARY OUTCOMES:
Event-free survival per independent review committee assessment | Up to 60 months

SECONDARY OUTCOMES:
Progression-free survival per independent review committee assessment | Up to 60 months
Overall survival | Up to 60 months
Incidence and severity of adverse events and their relationship to cemacabtagene ansegedleucel and ALLO-647 | Up to 60 months
  Adverse events, treatment emergent adverse events, serious adverse events, and adverse events of special interest evaluated by the investigator based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CRS and ICANS will be graded using ASTCT.
Incidence and severity of laboratory toxicities related to cemacabtagene ansegedleucel and ALLO-647 | Up to 60 months
  Change from baseline value and NCI toxicity grading of laboratory values outside of normal ranges using CTCAE version 5.0.
Minimal residual disease clearance | Up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Allogene Study Director, Study Director — Allogene Therapeutics, Inc.
Locations (59):
- United States (55):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Genesis Cancer and Blood Institute, Hot Springs, Arkansas
  - Alta Bates Summit Medical Center, Berkeley, California
  - City of Hope, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Advent Health Cancer Institute, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Augusta University Georgia Cancer Center, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - The University of Kansas Hospital, Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville Health Brown Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Missouri - Ellis Fischel Cancer Center, Columbia, Missouri
  - MidAmerica Cancer Care, Kansas City, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Astera Cancer Care, East Brunswick, New Jersey
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University Irving Medical Center and New York-Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Novant Health Cancer Institute- Hematology, Charlotte, North Carolina
  - Duke Blood Cancer Center, Durham, North Carolina
  - Oncology Hematology Care - Kenwood, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - Central South, Austin, Texas
  - Texas Oncology - Dallas Fort Worth, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Intermountain Health LDS Hospital, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Canada (4):
  - Arthur JE Child Comprehensive Cancer Centre, Calgary, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre - University Health Network, Toronto, Ontario
  - Hopital de'L'Enfant-Jesus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No